CLINICAL TRIAL: NCT05020223
Title: Comparison of Sucess of Pulpotomy, Direct Pulp Capping and Indirect Pulp Capping Modalities Using MTA in Primary Teeth (2 Years Follow up)
Brief Title: Comparison of Sucess of Pulpotomy, Direct Pulp Capping and Indirect Pulp Capping Modalities Using MTA in Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 601
Record Dates: First submitted 2021-08-15; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Deep Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MTA pulpotomy (Experimental): Usuing MTA as capping material for cervical pulpotomy as a treatment option for deep carious primary teeth with signs and symptoms of reversible pulpitis in presence of pulp exposure
  Interventions: Other: Vital pulp therapy
- MTA direct pulp capping (Experimental): Using MTA as capping material in case of trearment of deep carious primary teeth with signs and symptoms of reversible pulpitis with presence of pulp exposure
  Interventions: Other: Vital pulp therapy
- MTA indirect pulp capping (Experimental): Using MTA as indirect capping material for treatment of deep carious primary teeth with signs and symptoms of reversible pulpitis
  Interventions: Other: Vital pulp therapy

INTERVENTIONS:
Other: Vital pulp therapy — Vital pulp therapy different modalities for management of deep carious lesion in primary teeth

SUMMARY:
450 healthy children with primary teeth of deep carious lesions without signs or symptomes of irreverisible pulp damage was selected randompy divoded into 3 groups each of 150 children that inder go vital pulp therapy through pulpotomy,direct pulp capping or indirect pulp capping using MTA as capping material for each modality then followed up for 2 years or more

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Aged from 3 to 10 years old
* Deep cariuos primary tooth

Exclusion Criteria:

* Primary teeth with any signs or syptoms of irreversible pulpitis
* Primary teeth of any signs or symptomes of vitality loss
* Primary teeth near to exfoliation

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Tenderness | 2 years
  Precence or abscence
Abcess | 2 years
  Precence or abscence
Fistula | 2 years
  Precence or abscence
lamina dura | 2 years
  Intact or distorted
Periapical radiographic radiolucency | 2 years
  Precence or abcencs

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt